CLINICAL TRIAL: NCT03489044
Title: An Investigation of Levetiracetam in Alzheimer's Disease (ILiAD): a Proof of Concept Study
Brief Title: An Investigation of Levetiracetam in Alzheimer's Disease
Acronym: ILiAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other); Oxford Health NHS Foundation Trust (Other Government); Northumberland, Tyne and Wear NHS Foundation Trust (Other); UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRAS 203849; 2016-003109-32 (EudraCT Number)
Record Dates: First submitted 2018-03-09; First posted 2018-04-05 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Alzheimer Disease; Epilepsy
Keywords: Alzheimer; Seizure; Epilepsy; Anti-epileptic drug; Levetiracetam
MeSH Terms: conditions — Alzheimer Disease; Epilepsy; Seizures | interventions — Levetiracetam

STUDY DESIGN:
Intervention Model Description: Placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind, block randomised,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment arm (Levetiracetam) (Experimental): When in the active arm, after a baseline visit, participants will up-titrate Levetiracetam in 250mg steps at intervals of one week to Levetiracetam 500mg twice daily (two tablets twice daily). Participants will be maintained on Levetiracetam 500mg bd for four weeks and have a further full assessment at 8 weeks after being on Levetiracetam. Participants will then down-titrate Levetiracetam by 250mg every week until weaned to nil.
  Interventions: Drug: Levetiracetam
- Control arm (placebo oral tablets) (Placebo Comparator): When in the control arm, after a baseline visit, participants will up-titrate placebo (manufactured to look identical to Levetiracetam 250mg) in one tablet steps at intervals of one week to two tablets twice daily. Participants will be maintained on placebo for four weeks and have a further full assessment at 8 weeks after being on placebo. Participants will then down-titrate placebo by one tablet every week until weaned to nil.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Levetiracetam — To up-titrate Levetiracetam to 500mg (two tablets) twice daily followed by maintenance on Levetiracetam 500mg twice daily for four weeks and then down-titrate to nil over four weeks
  Arms: Active treatment arm (Levetiracetam)
Drug: Placebo Oral Tablet — To up-titrate placebo to two tablets twice daily followed by maintenance on placebo two tablets twice daily for four weeks and then down-titrate to nil over four weeks
  Arms: Control arm (placebo oral tablets)

SUMMARY:
The study proposed aims to evaluate the effect of Levetiracetam in patients with Alzheimer's disease (AD) in a Phase 2 Clinical Trial.

Levetiracetam is an established anti-epileptic medication that has been approved by NICE (UK) as a first line treatment for focal epilepsy. Levetiracetam is now generic and acts, as all anti-epileptic medications do, by stabilising neuronal networks. However, Levetiracetam appears unique amongst the anti-epileptic medications in being able to stabilise aberrant neuronal networks in Alzheimer's disease. In both animal models of AD and in patients with mild cognitive impairment, Levetiracetam can offer benefit to cognition.

The investigators therefore aim to test whether Levetiracetam, through stabilisation of neuronal networks, may offer benefit to cognition in patients with AD.

DETAILED DESCRIPTION:
Lay Summary:

Alzheimer's disease affects around 800,000 people in the UK alone and costs almost £23 billion per year. The only currently licensed treatments for Alzheimer's disease offer modest benefit at best. Seizures are more common in people with Alzheimer's disease and people with Alzheimer's disease may also have evidence of abnormal brainwave activity without having obvious seizures. Seizures may contribute to the loss of nerve cells and abnormal brainwave activity can disrupt thinking and memory. This abnormal electrical activity is therefore a potentially important drug target.

The anti-epileptic drug Levetiracetam can reduce abnormal brainwave activity and reverse memory deficits in a mouse model of Alzheimer's disease. Levetiracetam can also improve memory difficulties seen in people with mild cognitive impairment, a pre-cursor to Alzheimer's disease. Clinical use of Levetiracetam is already widespread and it is recommended by The National Institute of Health and Care Excellence as a first line treatment for seizures. Levetiracetam is generic (off-patent), is not known to interact with any other drugs and is well tolerated. A promising, cheap and safe approach might be to use Levetiracetam as a treatment to help with memory difficulties in Alzheimer's disease.

The proposed project is a proof of concept study. The investigators wish to allocate thirty patients with Alzheimer's disease with no history of previous seizure to initially receive either Levetiracetam or placebo before patients 'cross-over' so that the participants who initially received Levetiracetam are then given placebo and vice-versa. The effect that Levetiracetam has on memory in Alzheimer's disease will be studied using several standardised scales. Tests that the investigators have developed to better detect subtle improvements in thinking will also be used. Patients will have a straightforward, non-invasive test called an electroencephalogram to look at their brainwave activity at the start of the study, as there may be brainwave markers that might help to predict which patients would benefit most from Levetiracetam.

This study evaluates if an anti-epileptic medication can offer meaningful benefit to patients with Alzheimer's disease. If this study is successful, the next step will be to rapidly progress to a larger study to establish whether Levetiracetam may be a useful and cost-effective treatment for patients with Alzheimer's disease.

Main hypothesis:

1. Treatment with the anti-epileptic drug Levetiracetam will be of benefit to cognitive deficits in Alzheimer's disease because electrophysiological disruption of neuronal networks contributes to the pathophysiology of the condition.
2. Treatment with Levetiracetam at a dose that is routinely utilized in older people with epilepsy will be well tolerated in patients with Alzheimer's disease and, in particular, will not adversely affect mood
3. Electroencephalography (EEG) may offer a biomarker to predict which patients with Alzheimer's disease might be especially suited to treatment with Levetiracetam

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, 50 years or above.
* Diagnosed with mild to moderate AD (MMSE 10 to 26)
* Meets the National Institute of Aging-Alzheimer's Association criteria for probable AD (2011)
* Stable dose of current regular medication, including acetylcholinesterase inhibitors if applicable, for at least 4 weeks prior to trial entry.
* Female participants of child bearing potential and male participants whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the trial and for 3 months thereafter. Acceptable forms of contraception include: established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device (IUD) or intrauterine system (IUS); total abdominal hysterectomy; barrier methods of contraception (condom or occlusive cap with spermicide); male sterilisation, if the vasectomised partner is the sole partner for the subject; true abstinence, when this is in line with the preferred and usual lifestyle of the subject (periodic abstinence and withdrawal are not acceptable methods of contraception).
* Participant has clinically acceptable blood and urine test results (creatinine clearance >75 ml/minute; liver function tests <2x upper limit of normal) and ECG that does not demonstrate conduction block or significant ischaemia within three months of enrolment.
* In the Investigator's opinion, is able and willing to comply with all trial requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the trial.
* Reliable carer willing and available to assist with medication administration as well as to accompany participants during any home visits.

Exclusion Criteria:

* Pre-existing diagnosis of epilepsy
* Clinical or laboratory evidence of a cause other than AD as a cause of their dementia
* Laboratory evidence of significant renal impairment (creatinine clearance <75 ml/minute) or liver dysfunction (liver function tests >2x upper limit of normal) within the preceding three months
* Visual or motor impairment that investigator deems severe enough to impair ability to complete computerised based touch screen task
* Use of anti-epileptic medication for any indication (epilepsy, pain or migraine) within previous three months
* Other severe neurological or medical condition. Examples include, significant stroke, heart failure, chronic renal failure, chronic liver failure within last 3 months
* Major depression or other significant behavioural disturbance
* Known allergy to Levetiracetam or history of previous adverse reaction to Levetiracetam
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial.
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
* Participant with life expectancy of less than 6 months, or is inappropriate for placebo medication.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participants who have participated in another research trial involving an investigational medicinal product in the past 12 weeks Carer of participant with AD
* Carer has significant medical illness that will preclude adequate data capture during the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-10-28 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Effect of Levetiracetam on hippocampal function in patients with Alzheimer's disease as assessed by a computerised test of hippocampal binding | 18 months
  Change from baseline in measures of hippocampal binding on a standardised computer based test. Participants will be shown fractals on a screen, followed by a blank screen. The participants will be then shown one of the fractals they saw previously and a foil. The participants will have to identify which of the fractals they saw initially and then drag that fractal on the screen to the location where it appeared before. The computer will assess whether the participant correctly identifies which fractal had been seen previously and also assess how accurately the participant remembers the location of the previously shown fractal. The investigators will then evaluate whether there are any changes in the accuracy of remembering fractals/fractal position after exposure to Levetiracetam/placebo

SECONDARY OUTCOMES:
Number of participants with treatment related serious adverse events as reported on the serious adverse events proforma | 18 months
  To determine if use of Levetiracetam associates with significant side effects in patients with AD that have not experienced an overt seizure
Effect of Levetiracetam on mood in patients with Alzheimer's disease | 18 months
  Number of participants reporting change from baseline on the Neuropsychiatric Inventory
Effect of Levetiracetam on quality of life in patients with Alzheimer's disease as assessed by their principal carer | 18 months
  Number of participants with a change from baseline on Dementia Severity Rating Scale
Effect of Levetiracetam on quality of life in patients with Alzheimer's disease | 18 months
  Number of participants with a change from baseline on the Euro-QoL (EQ5D) measure
Determining role of the electroencephalogram in patients with Alzheimer's disease | 18 months
  Correlation of electroencephalogram recording with effect of Levetiracetam on cognition as assessed by a computer based test of hippocampal binding

CONTACTS AND LOCATIONS:
Overall Officials: Arjune Sen, PhD, FRCPE, Study Director — Nuffield Department of Clinical Neurosciences
Locations (1):
- Nuffield Department of Clinical Neuroscience, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
It is possible that irretrievably anonymised data will be shared with other researchers dependent on securing relevant ethical approval

REFERENCES:
- [Derived] Sen A, Akinola M, Tai XY, Symmonds M, Davis Jones G, Mura S, Galloway J, Hallam A, Chan JYC, Koychev I, Butler C, Geddes J, Van Der Putt R, Thompson S, Manohar SG, Frangou E, Love S, McShane R, Husain M. An Investigation of Levetiracetam in Alzheimer's Disease (ILiAD): a double-blind, placebo-controlled, randomised crossover proof of concept study. Trials. 2021 Jul 31;22(1):508. doi: 10.1186/s13063-021-05404-4. PMID 34332638
- [Derived] Liu J, Wang LN. Treatment of epilepsy for people with Alzheimer's disease. Cochrane Database Syst Rev. 2021 May 11;5(5):CD011922. doi: 10.1002/14651858.CD011922.pub4. PMID 33973646